CLINICAL TRIAL: NCT06115850
Title: Effect of Music Intervention on Anxiety in Cancer Patients Undergoing Initial Radiation Therapy: A Randomized Clinical Trial
Brief Title: Effect of Music Intervention on Anxiety in Cancer Patients Undergoing Initial Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-a-037
Record Dates: First submitted 2023-10-26; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-01

CONDITIONS: Cancer Patients; Anxiety; Music Intervention; Radiation Therapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Music intervention (No Intervention): Anxiety assessment questionnaires were administered before the treatment began and after 2 weeks of treatment. Physiological parameters, including heart rate, systolic and diastolic blood pressure, and blood oxygen levels, were monitored before and after 2 weeks of treatment.
- Music intervention (Experimental): Anxiety assessment questionnaires were administered before the treatment began and after 2 weeks of treatment. Physiological parameters, including heart rate, systolic and diastolic blood pressure, and blood oxygen levels, were monitored before and after 2 weeks of treatment.
  Interventions: Procedure: Music

INTERVENTIONS:
Procedure: Music — In the music intervention group, the patients received music intervention during RT for 10 consecutive days and listened to music for approximately 10-15 minutes in each session.
  Arms: Music intervention

SUMMARY:
This prospective randomized trial evaluated the effect of music interventions on anxiety and nervousness during 10 consecutive days in individuals undergoing their first radiation therapy session.

DETAILED DESCRIPTION:
A total of 100 participants were enrolled and randomly assigned to either the music group or nonmusic group (n = 50 each). Investigators ensured an equal distribution of men and women, without considering the cancer type. To minimize confounding factors and prevent shared learning experiences or communication between the two groups, the participants in the experimental and control groups were scheduled for treatment at different times throughout the year (from January 1, 2022 to December 31, 2022). Anxiety assessment questionnaires were administered before the treatment began and after 2 weeks of treatment. Physiological parameters, including heart rate, systolic and diastolic blood pressure, and blood oxygen levels, were monitored before and after 2 weeks of treatment. In the music intervention group, the patients received music intervention during RT for 10 consecutive days and listened to music for approximately 10-15 minutes in each session. The music period was then followed by a 10-day period without music during treatment to evaluate the differences in the same individuals. In contrast, the control group did not receive music intervention throughout their entire RT period. Investigators observed the music intervention group for 2 weeks to ascertain any differences.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing RT for cancer for the first time
* patients with clear consciousness and normal hearing
* patients willing to respond to the questionnaire after the research process and purpose were explained to them.

Exclusion Criteria:

* patients who had previously undergone RT
* patients with diminished mental capacity or inability to satisfactorily participate in this study
* patients with moderate to severe hearing impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The physiological indicators - Heart rate | monitored before and after 2 weeks of treatment.
  Heart rate (Beat per minute ) were measured by a PHILIPS M1205A noninvasive physiological monitor.
The physiological indicators - Blood pressure | monitored before and after 2 weeks of treatment.
  Blood pressure (mmHg) were measured by a PHILIPS M1205A noninvasive physiological monitor.
The physiological indicators - Blood oxygen | monitored before and after 2 weeks of treatment.
  Blood oxygen (oxygen saturation，SO2 %) were measured by a PHILIPS M1205A noninvasive physiological monitor.
The anxiety status - Distress Thermometer | monitored before and after 2 weeks of treatment.
  Distress Thermometer (DT) which screens for psychological distress in patients with cancer as recommended by the National Comprehensive Cancer Network® (NCCN)
The anxiety status - Brief Symptom Rating Scale (BSRS-5) | monitored before and after 2 weeks of treatment.
  Brief Symptom Rating Scale (BSRS-5) or "Mood Thermometer," a 5-point Likert scale for assessing symptoms of emotional distress over 1 week. The total score ranges from 0 to 20.
The anxiety status - Beck Anxiety Inventory (BAI-C) | monitored before and after 2 weeks of treatment.
  Beck Anxiety Inventory (BAI-C, a 21-item self-reported questionnaire to assess anxiety symptoms on a 4-point scale, which has shown excellent internal consistency and test-retest reliability).
The anxiety status - Symptom Distress Thermometer (SDT) | monitored before and after 2 weeks of treatment.
  Symptom Distress Thermometer (SDT), a 10-point scale by the NCCN to evaluate distress levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan (r.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No